CLINICAL TRIAL: NCT06898346
Title: Maternal Health, Literacy and Pregnancy Outcomes: The Role of Specialized Nutrition Education
Brief Title: Ghana MHL Project, Tamale
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Ghana (Other); Nestlé Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000038987
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy
Keywords: Maternal Health Literacy; Dietary Diversity; Nutrition Education; RCT; Ghana; Nutrition Knowledge
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The treatment group will receive 6 nutrition education and counseling sessions
  Interventions: Behavioral: Nutrition Education
- Control (No Intervention): The control group will not receive the program's nutrition education intervention, However, to minimize the Hawthorne effect (Sedgwick, 2012) on the intervention, the control group will be visited as well but will receive education on personal hygiene only. All participants will continue to receive any education that is part of standard care from their primary care providers

INTERVENTIONS:
Behavioral: Nutrition Education — The treatment group will receive nutrition education (NE) and counseling 6 times. The 1st and 6th counselling sessions will be administered by a Registerd Dietitan in a health facility (weeks 21-22 and weeks 31-32). Four (4) bi-weekly follow-ups between these 2 sessions will be administered by Field Assistants (weeks 23, 25, 27 and 29) at the participant's home. NE will focus on dietary diversity and minimum meal frequency (Daniel et al, 2016; Gyimah et al., 2021), protein and energy intakes (Ota et al, 2015), intake of iron-rich foods (Otoo and Adam, 2016), guidelines for pregnancy with an emphasis on appropriate weight gain (Abubakar et al, 2016), and appropriate ingredients and food preparation methods required to optimize nutrition.
  Arms: Intervention

SUMMARY:
This study is designed to test a nutrition education program that focuses on local foods in northern Ghana. The goal is to help pregnant women eat a wider variety of foods, increase their intake of protein, energy, and iron-rich foods, and support healthy weight gain during pregnancy. We want to understand how this program impacts mothers' knowledge about nutrition and health, and how it affects the health of their babies. The program was created with input from pregnant women and health professionals in the community.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous pregnant (first-time) mothers (BMI<20kg/m2) between the ages of 18 and 40 attending antenatal sessions and in their second trimester, gestational ages (GA) of 16 weeks to 20 weeks, who are not carrying multiple fetuses

Exclusion Criteria:

* Women with pregnancies greater than 20 weeks gestation, to ensure adequate exposure to the intervention; mothers presenting with significant morbidity or who are admitted due to complications and mothers who cannot confirm an address or contact information and do not plan to deliver at a health facility as well as those who indicate that they would not deliver in the study region (those who will be out of town at time of delivery).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Health Literacy | 10-12 weeks
  Health literacy (HL) in women will be assessed using the All Aspects of Health Literacy Scale (AAHLS) developed by Chinn and McCarthy (2013), and maternal health literacy (MHL) will be assessed using an abridged version of the Maternal Health Literacy Inventory In Pregnancy (MHELIP) (Taheri et al, 2020).
Dietary Diversity in Women | 15-17 weeks
  Maternal dietary diversity will also be determined from 24-hr recalls by assessing how many food groups a woman consumed each day based on FAO definitions (FAO and FHI 360, 2016)

SECONDARY OUTCOMES:
Nutrition Knowledge | 15-17 weeks
  Maternal nutrition knowledge (NK) will be assessed with a questionnaire adapted from abridged versions of 2 previously validated questionnaires (de Jersey et al., 2013; Parmenter and Wardle, 1999)
Infant birth weight | 20 weeks
  Infant's weight at birth and other anthropometry (length, head circumference) is usually collected within 24 hours at the hospitals using infant weighing scales.

CONTACTS AND LOCATIONS:
Overall Officials: Ruthfirst EA Ayande, PhD, MSc, RD, Principal Investigator — Yale University; Gloria E Otoo, PhD, Principal Investigator — University of Ghana
Locations (1):
- Tamale Teaching Hospital, Tamale, Northern Region, Ghana

IPD SHARING:
Plan to Share IPD: No